CLINICAL TRIAL: NCT07387276
Title: "Effects of Multiple Muscle Recovery Techniques on Pain, Force, Temperature, and Muscle Oxygenation in Professional Athletes: A Randomized Crossover Trial"
Brief Title: "Recovery Techniques on Pain, Force and Muscle Oxygenation in Pro Athletes: A Crossover Trial"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 22
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Muscle Soreness; Delayed Onset Muscle Soreness; Athletic Injuries
Keywords: muscle recovery; SmO2; tecartherapy; shockwave therapy; massage
MeSH Terms: conditions — Myalgia; Athletic Injuries | interventions — Extracorporeal Shockwave Therapy; Manual Lymphatic Drainage; Cupping Therapy

STUDY DESIGN:
Intervention Model Description: "This is a randomized, 6-period, 6-sequence crossover clinical trial. Each participant will undergo six different recovery interventions (Shockwave Therapy, Percussion Massage, Manual Massage, TECAR Therapy, Cupping, and Pressotherapy) in a randomized order. To prevent carry-over effects, a minimum wash-out period of 1 week will be established between each intervention session. All participants will perform a standardized high-intensity effort to induce muscle fatigue prior to each recovery modality. Physiological and functional measurements (NIRS, thermography, algometry, and dynamometry) will be taken at baseline and immediately post-intervention in each period."
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the physical interventions (e.g., massage, shockwave therapy, cupping), participants and care providers cannot be blinded to the treatment assigned. However, to minimize bias, a double-blind approach will be implemented for data collection and analysis. The Outcomes Assessor (the person responsible for operating the Moxy NIRS monitors, algometer, and dynamometer) will be blinded to the specific recovery modality received by the athlete in each period. Furthermore, the statistical analysis will be performed by a blinded investigator using coded data to ensure objectivity in the comparison of the six recovery techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Extracorporeal Shockwave Therapy (ESWT) (Experimental): pplication of radial shockwave therapy using the Longest LGT-2500S device. A total of 2,000 pulses will be applied to the gastrocnemius muscle (medial and lateral heads) at a pressure of 2.5 bar and a frequency of 10-15 Hz. The intervention aims to improve local microcirculation and reduce myofascial stiffness.
  Interventions: Device: Extracorporeal Shockwave Therapy (ESWT)
- Percussive Therapy - Massage Gun (Experimental): Application of percussive massage using the Hyperice Hypervolt 2 Pro (commonly used in clinical studies). The intervention will last 5-10 minutes on the gastrocnemius at a frequency of 50 Hz (Level 3), focusing on the muscle-tendon junction to enhance neuromuscular recovery.
  Interventions: Device: Massage Gun
- TECAR Therapy - (Experimental): Use of the Fisiowarm 300 (Golden Star, Italy) diathermy system. The treatment will be applied for 15 minutes in a combination of capacitive and resistive modes at a frequency of 500 kHz. The intensity will be set to a thermal level (Type III) to promote deep vasodilation and metabolic clearance in the calf muscles.
  Interventions: Device: TECAR Therapy
- Expert Manual Sports Massage (Experimental): A 15-to-20-minute standardized sports massage session performed by a senior physiotherapist with over 20 years of experience in elite sports. The protocol includes deep effleurage, petrissage, and transverse friction to alleviate muscle tension and improve blood flow in the gastrocnemius.
  Interventions: Other: Manual Massage
- Intermittent Negative Pressure (Experimental): Application of intermittent negative pressure using the Physium System (multimodal vacuum therapy). The protocol consists of a 10-minute session on the gastrocnemius area to decompress tissue layers, enhance lymphatic drainage, and modulate mechanoreceptors for pain reduction.
  Interventions: Device: cupping
- Pressotherapy (Experimental): use of the Hermes professional pressotherapy system. The treatment will last 20 minutes with a sequential 6-chamber inflation cycle and a pressure of 70-80 mmHg, targeting the acceleration of venous return and reduction of post-effort edema.
  Interventions: Device: Pressotherapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy (ESWT) — Application of acoustic pulses to the gastrocnemius muscle to modulate tissue mechanotransduction and improve local microcirculation.
  Arms: Extracorporeal Shockwave Therapy (ESWT)
Device: Massage Gun — Mechanical vibration applied to the calf muscles to promote myofascial release and neuromuscular recovery through high-frequency percussion.
  Arms: Percussive Therapy - Massage Gun
Device: TECAR Therapy — Application of high-frequency electromagnetic energy (diathermy) to the lower limb to induce deep endogenous heat and accelerate metabolic waste removal.
  Arms: TECAR Therapy -
Other: Manual Massage — Systematic manipulation of soft tissues using manual techniques (effleurage and petrissage) focused on reducing muscle tension and perceived soreness.
  Arms: Expert Manual Sports Massage
Device: cupping — Controlled suction therapy applied to the gastrocnemius to create space between fascial layers and stimulate lymphatic and venous drainage.
  Arms: Intermittent Negative Pressure
Device: Pressotherapy — External pneumatic compression through a sequential inflation system to facilitate venous return and reduce lower limb edema post-effort.
  Arms: Pressotherapy

SUMMARY:
The goal of this clinical trial is to evaluate the impact of different passive post-effort recovery techniques on professional athletes. The main questions it aims to answer are:

-Do passive recovery modalities significantly improve muscle oxygenation and tissue temperature immediately after high-intensity effort? Which specific technique is most effective in reducing perceived pain (pressure pain threshold) and restoring muscle strength?

Researchers will compare six different therapeutic interventions-TECAR therapy, massage, intermittent negative pressure (cupping), shockwave therapy, percussion guns, and pressotherapy-to see which provides the superior immediate physiological and functional recovery effect. Participants will:

Perform a high-intensity physical effort designed to induce peripheral fatigue.Be randomly assigned to receive one of the six recovery protocols.Undergo objective measurements immediately after the intervention, including muscle oxygen saturation (NIRS), tissue thermography, algometry, and dynamometry.

DETAILED DESCRIPTION:
This project consists of a randomized, double-blind (tester and statistician), crossover clinical trial. The study aims to address the critical need for evidence-based recovery strategies in high-demand sports like basketball, where muscle overload is a primary risk factor for injuries.The investigation will focus on the immediate effects of six widely used physiotherapy modalities:

TECAR Therapy: Used to improve perfusion and modulate inflammation through deep tissue heating.

Percussive Massage (Massage Guns): Applied to reduce stiffness and enhance explosive force through mechanical vibration.

Shockwave Therapy (ESWT): Evaluated for its capacity to improve muscular microcirculation and accelerate tissue regeneration.

Pressotherapy (External Pneumatic Compression): Targeting the reduction of pain and the sensation of heaviness in the lower limbs.

Intermittent Negative Pressure (Cupping): Investigated for its role in improving blood flow and pain modulation Sports Massage: The traditional manual intervention for reducing delayed onset muscle soreness (DOMS) and improving flexibility. Physiological monitoring will be conducted using Near-Infrared Spectroscopy (NIRS) via Moxy Monitors to measure muscle oxygen saturation (SmO2) and total hemoglobin, providing direct data on muscle oxidative metabolism. Functional outcomes will be assessed through pressure pain thresholds (algometry) and isometric strength (dynamometry) to determine the effectiveness of each technique in restoring neuromuscular homeostasis.The study will be conducted at the Sierra Varona Physiotherapy Clinic (Toledo) between february and march 2026.

ELIGIBILITY:
Inclusion Criteria:

Professional or Semi-professional athletes (specifically basketball players or endurance athletes) with a minimum of 2 years of competitive experience.

Aged between 18 and 35 years.

Healthy individuals with no current musculoskeletal injuries in the lower limbs.

Regular training frequency of at least 4-5 sessions per week.

Signed informed consent to participate in the study and follow the 6-week crossover protocol.

Commitment to maintain similar nutritional and sleep habits throughout the duration of the study.

Exclusion Criteria:

Presence of any acute or chronic injury in the gastrocnemius or Achilles tendon in the last 6 months.

Contraindications for specific therapies:

For Shockwave Therapy: Blood clotting disorders or use of anticoagulants.

For TECAR/Diathermy: Metal implants in the lower limbs or pacemakers.

For Cupping: Acute skin infections or dermatological hypersensitivity.

Consumption of performance-enhancing drugs, anti-inflammatory medication (NSAIDs), or stimulants that could affect muscle oxygenation (SmO2) or pain perception.

Recent surgery in the lower extremities (within the last year).

Inability to complete the standardized fatigue protocol or attend all 6 intervention sessions.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
Muscle Oxygen Saturation (SmO2) | immediately post-effort (fatigue), and immediately post-intervention (recovery).
  Measured using Moxy Monitor (Near-Infrared Spectroscopy - NIRS). It evaluates the percentage of hemoglobin/myoglobin oxygenated in the gastrocnemius muscle.
Pressure Pain Threshold (PPT) | immediately post-effort (fatigue), and immediately post-intervention (recovery).
  Measured using a digital pressure algometer. It quantifies the minimum pressure (in kg/cm²) at which a participant perceives the stimulus as painful in the gastrocnemius.
Maximum Isometric Muscle Strength | immediately post-effort (fatigue), and immediately post-intervention (recovery).
  Measured using a handheld dynamometer. It evaluates the peak force (in Newtons) during a maximum voluntary isometric contraction of the calf muscles.

SECONDARY OUTCOMES:
Muscle Surface Temperature | immediately post-effort (fatigue), and immediately post-intervention (recovery).
  Measured using a digital infrared thermography camera. It assesses the changes in skin surface temperature over the gastrocnemius muscle area, reflecting changes in local blood flow.
Participant Satisfaction and Perceived Recovery | 5 minutes after each recovery intervention.
  Measured using a Visual Analog Scale (VAS) and a customized survey (Likert scale 1-5). Participants rate which recovery modality felt better and their perceived level of muscle readiness for a new effort.

IPD SHARING:
Plan to Share IPD: Yes
"De-identified individual participant data (including muscle oxygenation variables, pressure pain thresholds, and isometric strength values) will be made available upon reasonable request to the principal investigator. Data will be shared to facilitate meta-analyses or to verify the findings of this study, provided that the requesting researcher provides a methodologically sound proposal and signs a data use agreement to ensure athlete confidentiality."